CLINICAL TRIAL: NCT07146048
Title: A Non-Inferiority Trial of Stopping Penicillin in Early Rheumatic Heart Disease: GOAL-Stop
Acronym: GOAL-Stop
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Uganda Heart Institute (Other); Open Philanthropy (Other); Thrasher Research Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-0604
Record Dates: First submitted 2025-08-20; First posted 2025-08-28 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Rheumatic Heart Disease
Keywords: Rheumatic heart disease; global health; secondary prophylaxis; children
MeSH Terms: conditions — Rheumatic Heart Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Cardiologists who make up the adjudication panel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stop prophylaxis (No Intervention): The intervention arm will not receive prophylaxis.
- Continue prophylaxis (Active Comparator): The control arm will receive intramuscular benzathine benzylpenicillin G (BPG) prophylaxis (600,000 IU for children <30kg, 1.2 million IU for children ≥30kg), every 28 days for a 2-year period. The standard of care for RHD is BPG injections which is why the control arm is continuation of monthly injections.
  Interventions: Drug: Secondary Prophylaxis

INTERVENTIONS:
Drug: Secondary Prophylaxis — Continue standard of care with continued secondary antibiotic prophylaxis
  Arms: Continue prophylaxis

SUMMARY:
GOAL-Stop is a randomized, controlled, non-inferiority trial designed to evaluate whether discontinuing secondary antibiotic prophylaxis (SAP) is non-inferior to continuing SAP in preventing progression of rheumatic heart disease (RHD) among children and adolescents. The trial will enroll participants aged 5-20 years with previously diagnosed mild RHD who have received at least 2 years of SAP and who demonstrate either echocardiographic normalization or stability (persistent mild RHD). Participants will be randomized to either continue SAP or discontinue SAP for 2 years. The primary outcome is echocardiographic progression of RHD at 2 years, assessed by blinded adjudicators using the 2023 World Heart Federation criteria. Subgroup analyses will evaluate outcomes in participants with echocardiographic normalization versus stable mild RHD, and an exploratory analysis will assess whether outcomes differ by prior prophylaxis route (oral vs. intramuscular).

ELIGIBILITY:
Inclusion Criteria:

* Participated in GOALIE
* Concluded GOALIE with either echocardiographic normalization or stable mild RHD
* Between ages 5-20 years at time of enrollment

Exclusion Criteria:

* RHD Stage C/D at GOALIE end of study echocardiogram
* Relocation to extremely distant residence or school
* Clinically documented penicillin allergy

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 922 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-02-20 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence of echocardiographic progression of RHD at two years | Enrollment to the end of treatment at 2 years
  The Primary Outcome will be the presence of echocardiographic progression of RHD at two years, defined by the 2023 World Heart Federation Criteria (none, mild RHD (stage A/B), or moderate/severe RHD (stage C/D).

SECONDARY OUTCOMES:
Non-inferiority among sub-groups | Enrollment to the end of 2 years participation
  Number of participants who show echocardiographic progression (2023 World Heart Federation Criteria) between those with echocardiographic normalization and those with stabilized mild RHD

OTHER OUTCOMES:
Exploratory sub-analysis | enrollment to the end of 2 years of participation
  Number of echocardiographic progression outcomes based on the initial type of prophylaxis during the GOALIE Trial, oral prophylaxis vs. intramuscular prophylaxis.

IPD SHARING:
Plan to Share IPD: Undecided
Pending approval of consent form

REFERENCES:
- See also: Related Info — https://www.rrcuganda.org/